CLINICAL TRIAL: NCT07018583
Title: The Effectiveness of Pharmacist's Counseling and Self-Management Application Program on Asthma Management Outcomes Among Asthma Patients at a Midwest Chain Pharmacy in Iowa, United States
Brief Title: Pharmacist Counseling & Self-Management Program for Asthma Patients in a Midwest Chain Pharmacy, USA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nakhon Ratchasim Rajabhat University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NRRU2025-001_DON
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Asthma Patients
Keywords: Pharmacist-led-intervention; Asthma management; Asthma awareness

STUDY DESIGN:
Intervention Model Description: This interventional study is structured around established counseling principles and self-management theory, consisting of six sequential stages: Initial Disclosure, Problem Assessment, Commitment to Action, Skill Enhancement, Monitoring, and Follow-up and Evaluation. These stages are delivered through both in-person pharmacist counseling and a dedicated mobile application. The intervention follows a repeated-measures design, with assessments conducted at 3 and 6 months after enrollment.
  Participants are randomly assigned to one of two groups:
  The intervention group receives pharmacist-led counseling integrated with a self-management mobile application program.
  The control group receives usual care, including standard pharmacy services, without additional digital or structured counseling support.
Who Masked: Participant
Masking Description: Outcome assessors and data analysts will be blinded to group assignments to minimize bias during data collection and statistical analysis. The researcher will not be blinded due to the nature of usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-Led Counseling and Self-Management App Program (Experimental): Participants in this arm will receive a structured asthma management intervention consisting of pharmacist-led counseling and access to the "Don R.Ph. Asthma Management Application."
  Interventions: Behavioral: Pharmacist's Counseling and Self-Management Application Program
- Comparator: Usual Care (Standard Pharmacy Services) (Active Comparator): The participants will recieve standard pharmacy practices such as medication reviews, patient education during the initial visit or when medication changes occur, and counseling upon patient request. No additional structured counseling or self-management tools are provided.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Pharmacist's Counseling and Self-Management Application Program — This interventional study is structured around established counseling principles and self-management theory, consisting of six sequential stages: Initial Disclosure, Problem Assessment, Commitment to Action, Skill Enhancement, Monitoring, and Follow-up and Evaluation. These stages are delivered through both in-person pharmacist counseling and a dedicated mobile application. The intervention follows a repeated-measures design, with assessments conducted at 3 and 6 months after enrollment.
  Arms: Pharmacist-Led Counseling and Self-Management App Program
Behavioral: Usual Care — Usual care or Standard pharmacy practices such as medication reviews, patient education during the initial visit or when medication changes occur, and counseling upon patient request. No additional structured counseling or self-management tools are provided.
  Arms: Comparator: Usual Care (Standard Pharmacy Services)

SUMMARY:
This clinical trial aims to evaluate the effectiveness of a pharmacist-led counseling and self-management application program on improving asthma management outcomes among adult patients with asthma receiving care at a Midwest chain pharmacy in Iowa, United States.

The study investigates whether integrating the pharmacist counseling with self-management theory can enhance patients' medication adherence, asthma control, inhaler technique, and overall asthma awareness. These outcomes will be assessed at both 3 and 6 months after enrollment.

Participants will be randomly assigned to one of two arms. The intervention group, which will receive a comprehensive pharmacist-led counseling program supported by a mobile application ("Don R.Ph Application").

The control group, which will receive standard pharmacy care as per usual practice.

DETAILED DESCRIPTION:
Protocol of the Study This research employs a randomized controlled trial (RCT) methodology to evaluate the effectiveness of a pharmacist-led counseling and self-management application program for asthma management.

Study Design:

This is a 6-month, repeated-measures, parallel-group RCT designed to assess the intervention's impact on asthma outcomes. The study comprises two groups:

Intervention Group: Participants will receive a pharmacist-led counseling session combined with access to a self-management mobile application.

Control Group: Participants will receive usual care provided within the pharmacy setting.

Data Collection Process:

1. Screening: Eligible participants will be identified based on predefined inclusion and exclusion criteria.
2. Randomization and Blinding: After screening, eligible participants will be randomly assigned to either the intervention or control group in a single-blind manner.

Sample Size and Allocation:

* A total of 397 patients with asthma diagnosis codes will be initially screened for eligibility.
* Among these, 220 patients meeting the criteria will be assigned unique codes and recorded in Microsoft Excel.

Using simple randomization, 42 participants will be allocated to each group, maintaining a 1:1 ratio via computerized random number generation (using the RANDBETWEEN function in Excel) to minimize selection bias.

4. Informed Consent: Participants will be provided with detailed study information and will give written informed consent prior to participation.

5. Baseline Data Collection: Baseline demographic and clinical data will be gathered for all participants in both groups.

6. Interventions:

* Intervention Group: Participants will undergo a structured pharmacist-led counseling and self-management program utilizing the "Don R.Ph. Asthma Management Application," a digital tool designed to support and monitor asthma management through six core steps over two 3-month cycles.
* Control Group: Participants will receive standard pharmacy care, including medication reviews, patient education, and counseling on medication use as needed or upon request.

  7. Follow-up and Duration: Follow-up data will be collected at three and six months during and after the intervention period.

The study spans six months, with the intervention structured into six steps:

Month 1:

Step 1: Initial Disclosure Step 2: Problem Assessment Step 3: Commitment to Action Step 4: Skill Enhancement

Month 2:

Step 5: Monitoring via mobile application

Month 3:

Step 6: Follow-up and evaluation via mobile app and in-person counseling

This cycle will be repeated in months 4-6 to reinforce behavioral changes and optimize long-term outcomes.

The "Don R.Ph. Asthma Management Application" is a digital platform to support and monitor the pharmacist-led counseling process through eight key features:

1. Setting Your Goal! - Enables patients to establish personalized asthma management objectives.
2. Understanding Asthma - Offers educational videos about asthma and proper medication use.
3. How to Use Inhalers - Demonstrates correct inhaler techniques via videos.
4. Healthy Lifestyle - Shares practical tips to promote overall health and asthma control.
5. Asthma Self-Management & Action Plan - Guides patients in creating and following tailored action plans.
6. Automated Consultation - Provides automated, personalized guidance and reminders
7. Let Us Know - Offers quick access to emergency pharmacist contact for urgent concerns.
8. Assess Your Goal Achievement - Allows patients to monitor their progress toward management goals through self-assessment tools.

ELIGIBILITY:
Inclusion criteria:

1. Adult patients with asthma are 25 - 64 years of age.
2. Have been receiving medications from the pharmacy of either Inhaled Corticosteroids (ICS) or a fixed combination of ICS with a long-acting beta-agonist (bronchodilator) and regular patronage of the pharmacy for the previous six months.
3. Confirmed diagnosis from either the physician's diagnosis or the patient's self-report.
4. No respiratory comorbidities (i.e., COPD or lung diseases).
5. Uses a smartphone (IOS or Android).
6. Ability to communicate with the pharmacist in English.
7. Volunteer to participate in the program for the period.

Exclusion criteria:

1. The adult patient with asthma aged < 25 years or > 64 years old.
2. The patient with one of the following - coronary heart disease, severe hypertension, severe heart failure, severe musculoskeletal disorder, mental health condition, dementia, chronic obstructive lung disease, or COVID-19.
3. Participating in another "Pharmacy Counseling or Education Program."
4. The patient does not have a smartphone (iOS or Android).
5. The patient does not have sufficient comprehension or the ability to communicate effectively in English.
6. The patient is unwilling or unable to participate in the entire program.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | Baseline, 3 months, and 6 months
  The Adherence to Asthma Medication Questionnaire (AAMQ-13) is a self-report scale developed by Nassar, Saini, Obeidat, and Basheti (2022). It consists of thirteen questions regarding the frequency of medication use, alterations, forgetfulness, and reasons for discontinuing medication over the past seven days. Each question is scored on a scale of 1 to 5, with options ranging from "Always, Often, Sometimes, Rarely, Never." The total score can range from 13 to 65.
  A low total score indicates a low level of medication adherence, while a high total score indicates a high level of medication adherence. However, the researcher conducted a statistical analysis to compare the mean medication adherence scores between the experimental and control groups after the intervention, and found a statistically significant difference.
Asthma Control | Baseline, 3 months, and 6 months
  The "Asthma Control Test (ACT)" is a self-administered questionnaire developed by Nathan (2004) to evaluate asthma control in patients. It consists of five questions that address asthma symptoms, medication use, and an overall assessment of asthma control over the past four weeks. Each question is scored on a scale of 1 to 5, with options ranging from "all of the time, most of the time, some of the time, a little of the time, " to " none of the time." The total score can range from 5 to 25, providing insight into the patient's level of asthma control.
  A low total score indicates a low level of asthma control, while a high total score indicates a high level of asthma control. However, the researcher conducted a statistical analysis to compare the mean asthma control scores between the experimental and control groups after the intervention, and found a statistically significant difference.

SECONDARY OUTCOMES:
Inhaler technique skill | Baseline, 3 months, and 6 months
  "The Metered-Dose Inhaler technique; MDIs" NHLBI (2021) is used to assess inhaler technique skills. The assessment comprises ten items on how to use the inhaler, including removing and shaking the cap, breathing out, actuating the inhaler, inhaling, holding breath, and waiting before repeating the second puff. The assessment comprises "Competent technique (C) and "Improvement requires (I)," with a total score ranging from 0 to 12.
  A low total score indicates a low level of inhaler technique skills, while a high total score indicates a high level of inhaler technique skills. However, the researcher conducted a statistical analysis to compare the mean inhaler technique skills scores between the experimental and control groups after the intervention, and found a statistically significant difference.
Asthma Awareness | Baseline, 3 months, 6 months
  The self-report on asthma awareness, developed by the researcher, includes perceptions of asthma severity, lifestyle factors, environmental management, prevention strategies, identification of triggers and early symptoms, medication adherence, correct inhaler use, readiness to follow an asthma action plan, and the importance of follow-up care. The total number of questions on asthma awareness consists of fifteen items. Each question is scored on a scale of 1 to 5 with options ranging from "Strongly disagree, Disagree, Neutral, Agree, and Strongly disagree." The total score can range from 15 to 75.
  A low total score indicates a low level of asthma awareness, while a high total score indicates a high level of asthma awareness. However, the researcher conducted a statistical analysis to compare the mean asthma awareness scores between the experimental and control groups after the intervention, and found a statistically significant difference.

IPD SHARING:
Plan to Share IPD: Yes
1. De-identified individual participant data related to the study's primary and secondary outcomes, including data on medication adherence, asthma control scores, inhaler technique performance, and asthma awareness assessments.
  2. Study protocol, statistical analysis plan, and informed consent form (de-identified and redacted as appropriate).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1. Data will be made available beginning 6 months after publication of the primary study results, or 12 months after the completion of the trial, whichever occurs first.
  2. The data will be available for at least 5 years following its release.
Access Criteria: Qualified researchers affiliated with academic institutions, public health organizations, or non-profit entities.
URL: https://www.nrru.ac.th